CLINICAL TRIAL: NCT03003117
Title: Effectiveness of an Early Intervention Aiming at Promoting Healthy Diet, Lifestyle and Growth of Children Living in Situation of Social Disadvantage : the prEgnanCy and eArly Childhood nutrItion triaL (ECAIL)
Brief Title: The prEgnanCy and eArly Childhood nutrItion triaL (ECAIL)
Acronym: ECAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Red Cross (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Lille (Other); Association Programme MALIN (Unknown); Société Française de Pédiatrie (Unknown); Association Française de Pédiatrie Ambulatoire (Unknown)
Responsible Party: Principal Investigator, Sandrine LIORET, Senior Research Fellow, PhD, Institut National de la Santé Et de la Recherche Médicale, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-A00849-38; n°CPP 03/010/2014 (Other: Comité de Protection des Personnes Nord-Ouest 1)
Record Dates: First submitted 2016-12-21; First posted 2016-12-26 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Diet; Growth; Infant; Physical Activity; Sedentary Behavior
Keywords: Infant; Diet; Growth; Breastfeeding; Complementary feeding; Pregnancy; Body mass index; Social disadvantage; Randomized controlled trial; Education; Food vouchers; Physical activity; Screen
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Program (Experimental): Experimental: Intervention Program
  Interventions: Behavioral: Experimental: Intervention Program
- Usual Care (Active Comparator): Active comparator: Usual Care
  Interventions: Behavioral: Active comparator: Usual Care

INTERVENTIONS:
Behavioral: Experimental: Intervention Program — The home based educational component from the 3rd trimester of pregnancy to when the child is aged 24 months seeks to build knowledge, skills and social support (social cognitive theory, anticipatory guidance) to the parents regarding feeding practices (focussing on breastfeeding and complementary feeding), and lifestyle behaviors, consistent with the French Nutrition and Health Program (PNNS) guidelines (component 1). Fresh fruit and vegetable baskets, kitchen utensils and cooking devices are made available at a reduced price from the 3rd trimester of pregnancy to when the toddler is aged 24 m (component 2), along with the provision of follow-on formula, baby and family food vouchers from 6 to 24 m (component 3).
  One home visit is scheduled during the 3rd trimester of pregnancy. Another visit will take place in the maternity ward after the child is born. Five further home visits will take place when the child is aged 3, 6, 12, 18 and 24 m.
  Arms: Intervention Program
Behavioral: Active comparator: Usual Care — Usual Care reflects the standard treatment currently provided within the frame of the French health care system. One home visit is scheduled during the 3rd trimester of pregnancy. Another visit will take place in the maternity ward after the child is born. Five further home visits will take place when the child is aged 3, 6, 12, 18 and 24 m. If nutritional questions are raised by parents, dieticians will restrict their responses based on the food guides of the PNNS.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial among 800 socially disadvantaged pregnant women and their families to test the effectiveness of a multi-component home visitation nutrition program, compared to usual care, in promoting healthy feeding practices, lifestyle behaviors and growth in young children.

DETAILED DESCRIPTION:
This randomized controlled trial will test an early home based multi-component intervention program designed to promote healthy feeding practices and lifestyle behaviors in socially disadvantaged pregnant women and their families. It first seeks to build knowledge, skills and social support regarding maternal diet and feeding practices (with a focus on breastfeeding and complementary feeding), and lifestyle behaviors, within the frame of the French Nutrition and Health Program (Programme National Nutrition Santé, PNNS) while accounting for the cultural background and barriers of the targeted population (component 1). It also involves fresh fruit and vegetable baskets, kitchen utensils and cooking devices, being made available at a reduced price from the 3rd trimester of pregnancy to when the toddler is aged 24 months (component 2), along with the provision of follow-on formula, baby and family food vouchers from 6 to 24 months (component 3). The intervention group (n=400) will benefit from these 3 program components. The control group (n=400) will receive usual care, restricted to general information on healthy eating provided by the food guides of the PNNS. The ECAIL study will assess the program's effectiveness on lifestyle behaviors and growth in the first 2 years of life.

Noteworthy, the program evaluated for effectiveness with the ECAIL trial is an existing program, called the MALIN program (https://www.programme-malin.com/), which has been progressively implemented in mainland France since 2012, to the exception of the ECAIL study area. Since 2019, counselling on movement behaviors, including the promotion of physical activity and the prevention of sedentary behaviors (e.g. screen time), has been added to the diet and feeding practices educational component; discount vouchers have further encompassed other healthy foods and products appropriate for all family members; and online sales for kitchen utensils and cooking devices have been started too.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman at her 3rd term of pregnancy
* Healthy
* Aged ≥ 18 years
* From a socially disadvantaged background
* Living in Lille, Lomme, Loos, Faches-Thumesnil, Ronchin, Hellemmes, Haubourdin, La Madeleine, Lambersart, Mons-en-Baroeul, Saint-André-Lez-Lille, Wattignies, Villeneuve-d'Ascq, Marcq-en-Barœul or Wasquehal; or in the Valenciennes conurbation.
* Willing and able to sign informed consent
* Who, in the Investigator's judgement, is able to comply with the protocol or study procedures (including French speaking)
* If twins are born from this pregnancy, only one will be randomly selected for inclusion

Exclusion Criteria:

* Pregnant woman under guardianship
* Participation in any other interventional clinical trial that is not compatible with the participation into the ECAIL study
* No permanent mailing address
* Housed in emergency accommodation centres, hotels, movable dwellings or homeless
* Planning to move outside the study area prior to the child's first birthday
* Serious illness during pregnancy that could interfere with optimal participation in the ECAIL study
* Hard drug consumption
* Multiple pregnancy (≥3 foetuses).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of vegetable consumption (times/day) at age 2 years | 2 years of age
  Measured at 2 years using a food frequency questionnaire

SECONDARY OUTCOMES:
Breastfeeding initiation rate | Up to 2 years of age
  Measured at different time points from birth to 2 y (scheduled at birth, 3 months, 6 months, 12 months, 18 months and 24 months of age) using questionnaires
Predominant and any breastfeeding durations | Up to 2 years of age
  Measured at different time points from birth to 2 y (scheduled at birth, 3 months, 6 months, 12 months, 18 months and 24 months of age) using questionnaires
Age at complementary feeding introduction | Up to 2 years of age
  Measured at different time points from birth to 2 y (scheduled at birth, 3 months, 6 months, 12 months, 18 months and 24 months of age) using questionnaires
Age at first introduction of processed (but not baby-specific) foods | Up to 2 years of age
  Measured at different time points from birth to 2 y (scheduled at birth, 3 months, 6 months, 12 months, 18 months and 24 months of age) using questionnaires
Frequency of vegetable consumption (times/day) at age 1 year | 1 year of age
  Measured at 1 year using a food frequency questionnaire
Dietary patterns at age 1 year | 1 year of age
  Measured at 1 year using a food frequency questionnaire
Lifestyle patterns at age 1 year | 1 year of age
  Measured at 1 year using dietary variables from the food frequency questionnaire; and movement behavioral variables (physical activity and sedentary behaviors) measured with a questionnaire. Lifestyle patterns will be derived using principal component analysis
Weight growth velocity over the six first months of life | Up to 6 months of age
  Weight measured at different time points from birth to 6 months of age
BMI at age 2 years | 2 years of age
  Weight, length and BMI measured at different time points from birth to 2 y
Proportion of children that are overweight or obese at age 2 years | 2 years of age
  Weight, length and BMI measured at different time points from birth to 2 y
Dietary patterns at age 2 years | 2 years of age
  Measured at 2 years using a food frequency questionnaire
Lifestyle patterns at age 2 years | 2 years of age
  Measured at 2 years using dietary variables from the food frequency questionnaire; and movement behavioral variables (physical activity and sedentary behaviors) measured with a questionnaire. Lifestyle patterns will be derived using principal component analysis
Weight growth curves from birth to 2 y | Up to 2 years of age
  Weight measured at different time points from birth to 2 y
Length growth curves from birth to 2 y | Up to 2 years of age
  Length measured at different time points from birth to 2 y
BMI curves from birth to 2 y | Up to 2 years of age
  BMI measured at different time points from birth to 2 y

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Lioret, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Delphine Ley, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - University Hospital, Lille
  - Valenciennes Hospital, Monaco Hospital maternity, Valenciennes

IPD SHARING:
Plan to Share IPD: No